CLINICAL TRIAL: NCT02315716
Title: Carfilzomib/Cyclophosphamide/Dexamethasone with Maintenance Carfilzomib in Untreated Transplant-eligible Patients with Symptomatic MM to Evaluate the Benefit of Upfront ASCT
Brief Title: Carfilzomib/Cyclophosphamide/Dexamethasone with Maintenance Carfilzomib in Multiple Myeloma
Acronym: Cardamon
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/12/0500; 2014-000506-35 (EudraCT Number)
Record Dates: First submitted 2014-12-03; First posted 2014-12-12 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Carfilzomib
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Consolidation with 4 cycles of CarCyDex (Experimental): Patients responding to induction treatment will receive 4 further cycles of Carfilzomib, Cyclophosphamide and Dexamethasone (CarCyDex) treatment followed by 18 months of maintenance carfilzomib
  Interventions: Drug: Consolidation with 4 cycles of CarCyDex
- Autologous Stem Cell Transplant (ASCT) (Active Comparator): Patients responding to induction treatment will receive a melphalan conditioned autologous stem cell transplant followed by 18 months of maintenance carfilzomib
  Interventions: Procedure: Autologous Stem Cell Transplant (ASCT)

INTERVENTIONS:
Procedure: Autologous Stem Cell Transplant (ASCT) — Randomisation to melphalan conditioned autologous stem cell transplant
  Arms: Autologous Stem Cell Transplant (ASCT)
Drug: Consolidation with 4 cycles of CarCyDex — Randomisation to 4 further cycles of Carfilzomib, Cyclophosphamide and Dexamethasone for responding patients following 4 cycles of induction chemotherapy
  Arms: Consolidation with 4 cycles of CarCyDex

SUMMARY:
The Cardamon trial is a phase 2 trial using the standard chemotherapy drugs cyclophosphamide and dexamethasone in combination with a new drug called Carfilzomib in patients with multiple myeloma.

DETAILED DESCRIPTION:
Multiple Myeloma is a cancer of the bone marrow and, for those patients that are young and fit enough, the disease is usually treated with chemotherapy (sometimes called induction chemotherapy) followed by a stem cell transplant using the patient's own stem cells (autograft or Autologous Stem Cell Transplant). Unfortunately almost all patients will experience a relapse at some point following this treatment. After relapse there are a number of treatment options but eventually the disease will become resistant to further therapy.

The use of an Autologous Stem Cell Transplant (or Transplant) after initial chemotherapy treatment has been shown in studies to increase the amount of time that patients are without symptoms of their myeloma before unfortunately their disease relapses. However, recently more effective induction chemotherapy regimens have been developed and patients treated with these new regimens are able to achieve higher and deeper responses than those previously treated on older regimens. Many also achieve complete or very good partial response, which was rare with the traditional chemotherapy regimens.

So, the investigators now do not know if giving patients an Autologous Stem Cell Transplant straight after their initial induction chemotherapy is the best thing to do. It may be that patients who respond well to a new drug containing regimen will obtain most benefit from their stem cells if these stem cells are frozen and stored, so that they can be used when their disease relapses.

In the Cardamon trial, the investigators will directly compare the outcome of patients who receive a transplant, versus those patients who do not and who instead receive Consolidation therapy. After induction treatment and stem cell harvest, patients will be randomly allocated to receive either a transplant or to receive consolidation therapy. Patients in the Cardamon trial will also be given maintenance treatment. This is treatment that is given on an ongoing basis, after the transplant or after the Consolidation therapy. The aim of maintenance treatment is to prolong disease response and delay the time to relapse.

In summary the purpose of the Cardamon study is:

1. to confirm the high response rate to a new treatment regime that includes Carfilzomib plus 2 standard chemotherapy drugs used for the treatment of Multiple Myeloma,
2. to investigate whether patients who respond well to this new Carfilzomib-containing induction regimen are able to maintain a long remission period without having an Autologous Stem Cell Transplant 'up-front', and
3. to find out if maintenance treatment with Carfilzomib is able to further reduce the number of remaining myeloma cells in the bone marrow, using the Minimal Residual Disease test.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with symptomatic MM (see appendix 3) eligible for stem cell transplantation, with the exception of the following treatments:

  * local radiotherapy to relieve bone pain and/or spinal cord compression
  * bisphosphonates
  * corticosteroids within the last 3 months. Within 14 days prior to study entry, the maximum permitted dose is 160mg (i.e. 4 days of Dexamethasone at 40mg, or equivalent), unless otherwise agreed by the TMG.
* Suitable for high dose therapy and ASCT
* Age ≥ 18 years
* Life expectancy ≥ 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2)
* Measurable disease as defined by one of the following:

  * Secretory myeloma: Monoclonal protein in the serum (≥10 g/L) or monoclonal light chain in the urine (Bence Jones protein ≥200mg/24hours), or serum free light chain (SFLC, involved light chain ≥100mg/L provided the FLC ratio is abnormal)
  * Non-secretory myeloma:
* Either ≥30% clonal plasma cells in bone marrow (aspirate or trephine)
* Or 10-30% clonal plasma cells in the marrow and >1 soft tissue or extra-osseous plasmacytoma ≥ 2 cm that is measurable for response assessment by CT or MRI
* Adequate hepatic function, with serum ALT ≤ 3.5 times the upper limit of normal and serum direct bilirubin ≤ 2 mg/dL (34 µmol/L) within 14 days prior to registration
* Absolute neutrophil count (ANC) ≥ 1.0 × 109/L within 14 days prior to registration and subject has not received any growth factor support within 7 days of testing. ANC≥0.8x109/L allowed for patients with racial neutropenia.
* Haemoglobin ≥ 8 g/dL (80 g/L) within 14 days prior to registration (subjects may be receiving red blood cell (RBC) transfusions in accordance with institutional guidelines)
* Platelet count ≥ 75 × 109/L (≥ 50 × 109/L if myeloma involvement in the bone marrow is > 50%) within 14 days prior to registration and subject has not received any platelet transfusions within 7 days prior to testing.
* Creatinine clearance (CrCl) ≥ 30 mL/minute within 14 days prior to registration, either measured or calculated using a standard formula (e.g. Cockcroft and Gault).
* Written informed consent
* Females of childbearing potential (FCBP) must agree to ongoing pregnancy testing and to practice contraception.
* Male subjects must agree to practice contraception.

Exclusion criteria

* Pregnant or breast-feeding females (lactating women may participate if breastfeeding ceases for the duration of trial treatment and until 12 months after last treatment)
* Previous systemic chemotherapy for myeloma, with the exception of steroids, as detailed above (see section 6.3.1)
* Any major surgery within 21 days prior to registration which in the investigator's opinion would compromise trial treatment and/or the patient's ability to comply with trial visits. Surgery to relieve spinal cord compression or for treatment of bone fractures is permitted.
* Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) 7 days prior to planned start of treatment, unless otherwise agreed by the TMG.
* Known human immunodeficiency virus (HIV) infection
* Active hepatitis B or C infection (refer to appendix 4)
* Unstable angina or myocardial infarction within 4 months prior to registration, NYHA Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to registration
* Non-haematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localised transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
* Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to registration
* Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilise carfilzomib)
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary, cardiac or renal impairment
* Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to registration
* Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Response rate | Within 4 weeks of the end of induction treatment
  Major response rate (sCR, CR & VGPR) to 4 cycles of CarCyDex
PFS | 2 years after randomisation
  Progression free survival at 2 years for both ASCT and non-ASCT (consolidation) arms

SECONDARY OUTCOMES:
To assess toxicity and tolerability of CarCyDex and carfilzomib as maintenance therapy in untreated patients with symptomatic multiple myeloma | From start of treatment until 30 days post end of maintenance treatment
  Adverse Events (including peripheral neuropathy), dose reductions and delays, tolerability of the induction and maintenance regimens (treatment delays, discontinuation rates)
Disease response rate | Within 4 weeks of the end of induction treatment
  Disease response rate (sCR, CR, VGPR, PR) to CarCyDex induction
PFS | Assessed every 6 months from the end of treatment until 36 months post induction
  PFS in both the ASCT and non-ASCT arms
Overall survival | Assessed every 6 months from the end of treatment until 36 months post induction
  Overall survival in both the ASCT and non-ASCT arms
MRD conversion following treatment | Baseline, Day 100 post ASCT or within 4 weeks of the end of consolidation treatment
  Improvement in disease response and conversion from MRD-positive to MRD-negative post ASCT and post Consolidation
MRD conversion following maintenance | Baseline, after 6 months of maintenance
  Improvement in disease response and conversion from MRD-positive to MRD-negative after 6 months of maintenance treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kwee Yong, Principal Investigator — University College, London
Locations (20):
- United Kingdom (20):
  - Queen's Hospital, Romford, Essex
  - Royal United Hospital, Bath
  - Birmingham Heartlands Hospital, Birmingham
  - NHS Lanarkshire, Bothwell
  - Bradford Royal Infirmary, Bradford
  - Kent and Canterbury Hospital, Canterbury
  - University Hospital of Wales, Cardiff
  - Medway NHS Foundation Trust, Gillingham
  - St James' Hospital, Leeds
  - St Bartholomew's Hospital, London
  - Barnet Hospital, London
  - Guy's Hospital, London
  - King's College Hospital, London
  - St George's Hospital, London
  - University College London Hospital, London
  - Maidstone and Tunbridge Wells, Maidstone
  - Churchill Hospital, Oxford
  - Royal Hallamshire Hospital, Sheffield
  - Royal Stoke University Hospital, Stoke
  - City Hospital Sunderland, Sunderland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yong K, Wilson W, de Tute RM, Camilleri M, Ramasamy K, Streetly M, Sive J, Bygrave CA, Benjamin R, Chapman M, Chavda SJ, Phillips EH, Del Mar Cuadrado M, Pang G, Jenner R, Dadaga T, Kamora S, Cavenagh J, Clifton-Hadley L, Owen RG, Popat R. Upfront autologous haematopoietic stem-cell transplantation versus carfilzomib-cyclophosphamide-dexamethasone consolidation with carfilzomib maintenance in patients with newly diagnosed multiple myeloma in England and Wales (CARDAMON): a randomised, phase 2, non-inferiority trial. Lancet Haematol. 2023 Feb;10(2):e93-e106. doi: 10.1016/S2352-3026(22)00350-7. Epub 2022 Dec 15. PMID 36529145